CLINICAL TRIAL: NCT00851123
Title: Modified Constrained - Induced Movement Therapy Compared to Intensive Bimanual Training for Subacute Stroke Patients. A Randomized Controlled Trial
Brief Title: Modified Constrained - Induced Movement Therapy Compared to Intensive Bimanual Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruitment difficulties the trial was stopped after an interim analysis at 30 patients.
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Principal Investigator, Iris Ch. Brunner, Research fellow, MSc, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UiB24126
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Stroke
Keywords: Stroke; arm paresis; mCIMT; bimanual training; rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Modified Constraint-Induced Movement therapy (Experimental): Modified Constraint-Induced Movement Therapy at the rehabilitation unit or in an outpatient clinic.
  Interventions: Behavioral: Modified Constraint-Induced Movement therapy
- 2.Task-specific bimanual training (Experimental): Task-specific bimanual training at the rehabilitation unit or in an outpatient clinic.
  Interventions: Behavioral: Task-specific bimanual training

INTERVENTIONS:
Behavioral: Modified Constraint-Induced Movement therapy — Four hours of treatment a week for four weeks by a physiotherapist or an occupational therapist emphasizing the affected arm. Patients will receive an individually tailored home training program and are supposed to train 2-3 hours daily on their own. A restraining mitt has to be worn 5 hours a day.
  Arms: 1. Modified Constraint-Induced Movement therapy
Behavioral: Task-specific bimanual training — Four hours of treatment a week for four weeks by a physiotherapist or an occupational therapist emphasizing bimanual tasks. Patients will receive an individually tailored home training program and are supposed to train 2-3 hours daily on their own.
  Arms: 2.Task-specific bimanual training

SUMMARY:
The purpose of the study is to evaluate the benefit of two different treatment approaches for the hemiplegic arm, modified Constraint-Induced Movement Therapy and task-related bimanual training.

DETAILED DESCRIPTION:
Detailed description:

Constrained-Induced Movement Therapy seems to be an efficacious treatment approach for a certain subgroup of patients with moderate to mild hemiparesis after stroke. Still it remains unclear whether the training intensity or restriction of the better arm plays the bigger role. CIMT or mCIMT is usually compared to standard care of lower intensity with no constraint of the better arm, or other treatments that do not focus on functional (task-specific) training for the hemiplegic arm. Bimanual training, implying training of activities requiring use of both arms, may however, be even more effective than mCIMT, provided that the training is of similar intensity. The purposes of this study are:

1. To compare the functional effect of mCIMT to bimanual training of equal intensity in order to examine if one of the treatment approaches is superior to the other regarding the regaining of motor abilities.
2. Based on fMRI scans of a subgroup of patients, to examine whether cortical reorganization after stroke differs depending on the type of treatment received (mCIMT vs bimanual training).
3. To examine the rationale for implementing new treatment approaches in primary- and secondary health care, and thereby contribute to improved coordination between specialist and municipal health care systems.

Patients in both groups will participate in a 4 week training program, either mCIMT or bimanual. In both groups cognitive techniques will be used to increase adherence. The patients will be examined when screening, before and after the intervention, and 3 months after completed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Upper extremity hemiparesis
* Between 2 and 16 weeks post-stroke
* At least 10º active extension of the wrist and at least 10º active extension of the thumb and at least 2 additional fingers

Exclusion Criteria:

* Cognitive problems, Mini Mental Status < 24
* Excessive pain in the paretic extremity
* Major medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Action Reach Arm Test | 3 years

SECONDARY OUTCOMES:
Motor Activity Log | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Iris C. Brunner, MSc, Principal Investigator — University of Bergen